CLINICAL TRIAL: NCT06867874
Title: Shedding of Syncytiotrophoblast-derived Extracellular Vesicles is Increased in Placenta Previa and Accreta Spectrum: a Case-control Study.
Brief Title: Syncytiotrophoblast-derived Extracellular Vesicles in Placenta Previa and Accreta Spectrum
Acronym: PAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5606
Record Dates: First submitted 2023-07-10; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-07

CONDITIONS: Placenta Previa; Placenta Accreta Spectrum
MeSH Terms: conditions — Placenta Previa; Placenta Accreta | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women with diagnosis of PP and PAS (Experimental): Pregnant women with abnormal placentation as placenta previa and accreta spectrum
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — Blood sample

SUMMARY:
The main goal of this case-control study is to quantify the levels of circulating syncytiotrophoblast-derived extracellular vesicles (STBEVs) in maternal blood in a population of women with placenta previa and placenta accreta spectrum.

DETAILED DESCRIPTION:
The main goal of this case-control study is to quantify the levels of circulating syncytiotrophoblast-derived extracellular vesicles (STBEVs) in maternal blood in a population of women with ultrasound diagnosis of PP with and without postpartum histopathologic diagnosis of PAS, compared to pregnant women with normal placentation.

The secondary aim of this case-control study is to characterize the multi-omics profiling of STBEVs cargo's (proteins, gene and transcripts) isolated from patients diagnosed with PP and PAS compared to the control population.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with diagnosis of placenta previa and accreta spectrum (cases)
* Healthy pregnant women
* > 18 years

Exclusion Criteria:

* < 18 years
* Twin pregnancies
* Chronic Infections
* Cancers
* Unable to give the written consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of circulating EVs from blood | 9 months (three trimester of pregnancy)
  Analysis of circulating syncytiotrophoblast-derived extracellular vesicles in the third trimester of pregnancy of women with abnormal placentation (placenta previa and placenta accreta spectrum)
Proteomics analysis of circulating EVs | 9 months (three trimester of pregnancy)
  Multi-omics profiling of circulating EVs cargo isolated from blood of pregnant women with abnormal placentation compared to healthy pregnant women

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Tersigni, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario A.Gemelli IRCSS, Roma, Italy